CLINICAL TRIAL: NCT02496910
Title: A Randomized,Open-label,Single Dose,Crossover Clinical Trial to Compare the Safety and Pharmacokinetics of YH22162 in Comparison to the Co-administration of Twynsta and Hygroton in Healthy Volunteers
Brief Title: PK Study of YH22162 FDC Compared to Combination of Twynsta and Hygroton
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: YH22162-102
Record Dates: First submitted 2015-06-30; First posted 2015-07-14 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 - Period 1 (Active Comparator): Telmisartan/Amlodipine 80/5 mg (FDC) and Chlorthalidone 25mg
  Interventions: Drug: Telmisartan/Amlodipine 80/5 mg (FDC); Drug: Chlorthalidone 25mg
- Group 2 - Period 1 (Experimental): YH22162 FDC tablet of Yuhan Corporation
  Interventions: Drug: YH22162
- Group 1 - Period 2 (Experimental): YH22162 FDC tablet of Yuhan Corporation
  Interventions: Drug: YH22162
- Group 2 - Period 2 (Active Comparator): Telmisartan/Amlodipine 80/5 mg (FDC) and Chlorthalidone 25mg
  Interventions: Drug: Telmisartan/Amlodipine 80/5 mg (FDC); Drug: Chlorthalidone 25mg

INTERVENTIONS:
Drug: YH22162
  Arms: Group 1 - Period 2; Group 2 - Period 1
Drug: Telmisartan/Amlodipine 80/5 mg (FDC)
  Other Names: Twinstar 80/5 mg
  Arms: Group 1 - Period 1; Group 2 - Period 2
Drug: Chlorthalidone 25mg
  Other Names: Hygroton 25mg
  Arms: Group 1 - Period 1; Group 2 - Period 2

SUMMARY:
This is a Randomized, open-label, single-dose, 2-treatment, 2-period, 2-sequence crossover design.

DETAILED DESCRIPTION:
This is a 2 by 2 cross-over study to evaluate pharmacokinetics of YH22162 FDC compared to reference twynsta and Hygroton co-administered in two groups enrolling healthy adult male subjects under fasting conditions.

Subjects will be admitted to the clinic in the evening before Day 1. All subjects will receive a single oral dose of YH22162 FDC or twynsta and Hygroton co-administered in the morning on Day 1. All the subjects will remain in the clinical unit until completion of all assessments on Day 2 including collection post-dose PK sample. Subjects will return to the clinic for pharmacokinetic samples at scheduled time. The two treatment periods will be separated by a washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female with a body mass index(BMI) between 18.5 and 25 kg/m2
2. Who has not suffered from clinically significant disease
3. Provision of signed written informed consent

Exclusion Criteria:

1. History of and clinically significant disease
2. A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs.
3. Administration of other investigational products within 3 months prior to the first dosing.
4. Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to reasons including laboratory test results, ECGs, or vital signs.
5. Sitting blood pressure meeting the following criteria at screening: 150 ≥ systolic blood pressure ≤100 (mmHg) and 100 ≥ diastolic blood pressure ≤ 60 (mmHg)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence study is based on Cmax and AUC parameters | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, MD, Ph.D, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea